CLINICAL TRIAL: NCT02826330
Title: Evidence of Abnormal Fecal Microbiota in Healthy Subjects at High Risk for Crohn's Disease: Family Studies and Relations With a Particular Genetic Profile and Serological. Comparison of Affected Individuals, Their Siblings and Healthy Controls.
Brief Title: Abnormal Fecal Microbiota in Healthy Subjects at High Risk for Crohn's Disease
Acronym: MAGIC
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2011_21; 2012-A00802-41 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-06-29; First posted 2016-07-11 (Estimated); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Crohn's Disease; Genetic Predisposition
Keywords: Crohn's Disease; Healthy relatives; Dysbiosis; Biomarkers
MeSH Terms: conditions — Crohn Disease; Genetic Predisposition to Disease; Dysbiosis | interventions — Biomarkers

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood, saliva, stools
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- case Crohn disease: 60 cases with Crohn's Disease
  Interventions: Other: biomarkers
- first relative healthy: 2 healthy relatives per CD case (total 120)
  Interventions: Other: biomarkers
- controls: 60 controls matched on gender and age with CD cases
  Interventions: Other: biomarkers

INTERVENTIONS:
Other: biomarkers — fecal microbiota analysis antibodies in serum and saliva DNA polymorphisms
  Other Names: Dysbiosis

SUMMARY:
Transversal multicentric French study on the microbiota in patients with Crohn's disease and their first degree healthy relatives The primary objective is the comparison of microbiota between patients with CD, healthy controls non genetically linked and first degree healthy relatives of patients with CD.

DETAILED DESCRIPTION:
Crohn's disease is a chronic inflammatory bowel disease associating flares and remission periods. Its etiology is unknown and there are no specific therapy. CD affects young patients and has a major impact on quality of life. There are few population-based studies and there are about 2.5 million affected patients in Europe and North America. From data from EPIMAD Registry the number of affected patients in France should be 200 000. The Crohn's disease pathogenesis is bad known; It coul be the results of the activation of the gastro-intestinal immune system toward gut microbiota in genetically susceptible hosts. In CD patients there is an important ecologic modification of the flora with an excess of Bacteroidetes and Proteobacteria and a decrease of anti inflammatory bacteria (Firmicutes). In ileum of CD patients a specific E Coli (adherent and invasive E Colo) is found in two thirds of cases.The presence of this AIEC seems to be associated to the variant NOD2 (results from our team in multiplex families).

In a family with at least 1 patient with CD, the healthy first degree relatives present a high risk (* 10) to also develop a CD.

The primary objective is the comparison of microbiota between patients with CD, healthy controls non genetically linked and first degree healthy relatives of patients with CD. The first endpoint is the Lachnospiraceae rates in each group.

The secondary objectives are :

1. the search for an association between bacterial dysbiosis and different genetic backgrounds in patients with CD, their first degree healthy relatives and controls.
2. the quantification of potential invasive bacteria with invasive properties (E. coli including adherent-invasive E. coli, Shigella, Salmonella, Yersinia, Campylobacter), and fecal fungal flora (Candida albicans, in particular) and their association with genetic and serological profiles in patients with CD, their healthy relatives and control subjects.
3. a study of environmental risk factors using a questionnaire to be submitted to CD patients, their healthy relatives and control subjects.

ELIGIBILITY:
Inclusion Criteria:

Patient with Crohn's disease

* Patient > 18 years old
* Having at least one first degree health relative
* OK to participate to the project

First degree healthy relatives

* specific clinical questionnaire and dosing fecal calprotectin to ensure the absence of inflammatory pathology.
* OK to participate to the project

Exclusion Criteria:

* Intestinal resection.
* Pregnant or breastfeeding woman.
* subject under guardianship
* subject does not speak French
* person unable to speak
* taking antibiotics or bowel preparation will push 6 weeks stool specimens, after cessation treatments.

Ages: 8 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Transversal multicentric French study on the microbiota in patients with Crohn's disease (n=60) and their first degree healthy relatives (n=120) and controls (n=60).
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2013-10-03 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-04-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Lachnospiraceae bacteria in stools within 3 groups | 1 YEAR
  After extraction DNA, microbiota will be studied via study of ribosomal DNA 16S using quantitative PCR and pyroséquençage

SECONDARY OUTCOMES:
Number of bacteria Firmicutes phylum (including Faecalibacterium prausnitzii and Clostridium Leptum) in stools within 3 groups | 1 year
  After extraction DNA, microbiota will be studied via study of ribosomal DNA 16S using quantitative PCR and pyroséquençage
Define different genetic and serologic backgrounds within 3 groups | 1 year
  Genetic analysis will include 380 genetic variants génétiques that will be genotyped including classic variants involved in CD: variants or mutations of NOD2, NOD1, IL23R, ATG16L1, DGL5, TNF, IL6, NFKB1... genes. Serological analysis will included anti-OmpC, anti-I2 and ASCA auto antibodies.
Quantify of bacteria with invasive properties (including AIEC) within 3 groups | 1 year
  Amplify bacterial DNA of Salmonella Typhi (amplification of ITS area specific of ARNr 16S-23S gene. For AIEC, using of qPCR methods based on chuA and yjaA genes.
Study of environmental risk factors within 3 groups | 1 year
  Specific questionnaire on environmental risk factors including vaccination, antibiotic use, ionfections, Home facilities and Diet befor the CD diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Gower-Rousseau, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (10):
- France (10):
  - Amiens University & Hospital, Amiens
  - cLERMONT fERRAND University Hospital, Clermont-Ferrand
  - APHP Kremlin Bicêtre, Le Kremlin-Bicêtre
  - CHRU,Hôpital Jeanne de Flandres, Lille
  - Hôpital Claude Huriez, CHRU, Lille
  - Nancy University Hospital, Nancy
  - Aphp Necker, Paris
  - APHP Robert Debré, Paris
  - Aphp St Antoine, Paris
  - Rouen University Hospital, Rouen

IPD SHARING:
Plan to Share IPD: Undecided